CLINICAL TRIAL: NCT01593631
Title: A Combination of Yoghurt Bacteria and Acid Lactase From Aspergillus Oryzae Improves Lactose Digestion in Lactose Malabsorbers More Reliably Than Preparations Containing Acid Lactase or Yoghurt Bacteria Alone
Brief Title: Acid Lactase in Combination With Yoghurt Bacteria for Improvement of Lactose Digestion in Lactose Malabsorbers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitacare Gmbh & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120506000
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Lactose Malabsorption
Keywords: lactose malabsorption; lactose intolerance; lactose digestion; lactose maldigestion; acid lactase; yoghurt bacteria
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 2 billion lyoph. yoghurt bacteria (Active Comparator)
  Interventions: Dietary Supplement: Lyoph. yoghurt bacteria
- 3300 FCC acid lactase (Active Comparator)
  Interventions: Dietary Supplement: Acid lactase
- 9000 FCC acid lactase (Active Comparator)
  Interventions: Dietary Supplement: Acid lactase
- Combination of Substances of arm 1 and 2 (Active Comparator)
  Interventions: Dietary Supplement: Acid lactase plus yoghurt bacteria
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Acid lactase — capsules cotaining 3300 FCC units of acid lactase
  Arms: 3300 FCC acid lactase
Dietary Supplement: Acid lactase — capsules containing 9000 FCC of acid lactase
  Arms: 9000 FCC acid lactase
Dietary Supplement: Lyoph. yoghurt bacteria — capsules containing 2 billion lyoph. yoghurt bacteria
  Arms: 2 billion lyoph. yoghurt bacteria
Dietary Supplement: Acid lactase plus yoghurt bacteria — Capsules containing 3300 FCC of acid lactase and 2 billion lyoph. yoghurt bacteria
  Arms: Combination of Substances of arm 1 and 2
Dietary Supplement: Placebo — Capsules containing di-calcium-phosphate
  Arms: Placebo

SUMMARY:
Fermented dairy products, especially real Yoghurt, are often tolerated better by lactose malabsorbers than unfermented dairy products. The intake of dietary supplements containing acid Lactase derived from Aspergillus oryzae with lactose containing foodstuffs is known to reduce/alleviate symptoms of lactose intolerance in lactose malabsorbers. The study aims to compare the effect of the intake of a combination of yoghurt bacteria and acid lactase to the effect of yogurt bacteria or acid lactase alone on the lactose digestion in lactose malabsorbers. It is hypothized that the combination preparation will be more effective and/or will show a more reliable effect than the two mono-preparations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of African or Asian origin.
* Older than 18 years
* Written informed consent

Exclusion Criteria:

* Participation in a clinical study with a drug or a medical product withing the last 30 days;
* Inability to comply with the study protocol;
* Allergy to milk protein;
* Intolerance against lactase preparations;
* Known metabolic or gastrointestinal diseases which affect the absorption, metabolism or excretion of food components except lactose maldigestion;
* Intake of drugs influencing resorption of food components or gastrointestinal motility;
* Surgery within the last three months which still affect the current status of health;
* Psychiatric diseases
* Epilepsia
* Risk for suicide
* Eating disorders, e.g. anorexia, bulimia
* Alcohol or drug abuse
* Legal incapacity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Increase in hydrogen concentration in the breath (H2-exhalation breath test) | Every 20 minutes for 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- tecura GmbH Medicine & Biotechnics - Dept. of Clinical Research, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] de Vrese M, Laue C, Offick B, Soeth E, Repenning F, Thoss A, Schrezenmeir J. A combination of acid lactase from Aspergillus oryzae and yogurt bacteria improves lactose digestion in lactose maldigesters synergistically: A randomized, controlled, double-blind cross-over trial. Clin Nutr. 2015 Jun;34(3):394-9. doi: 10.1016/j.clnu.2014.06.012. Epub 2014 Jul 8. PMID 25042846